CLINICAL TRIAL: NCT01209442
Title: A Pilot Phase II Trial of Hypofractionated Intensity-Modulated Radiation Therapy (Hypo-IMRT) Combining With Temozolomide (TMZ) and Bevacizumab for Patients With Newly Diagnosed Glioblastoma Multiforme (GBM)
Brief Title: Hypofractionated Intensity-Modulated Radiation Therapy With Temozolomide and Bevacizumab for Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-0274.cc; AVF4733s (Other Grant/Funding Number: Genentech, Inc)
Record Dates: First submitted 2010-09-23; First posted 2010-09-27 (Estimated); Results first posted 2019-04-12 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Glioblastoma Multiforme
Keywords: Glioblastoma; Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — Bevacizumab; Temozolomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RT with Temozolomide and Bevacizumab (Experimental): Patients will be treated with hypofractionated IMRT (60 Gy in 10 Fx) and daily TMZ at 75 mg/m2 qd concurrent with IMRT (including weekends and holidays). Bevacizumab will be administered at 10 mg/kg on day 1 and day 15. Day 1 and the 1st Fx of IMRT must start on the same day. Four to six weeks following completion of concurrent IMRT, TMZ and bevacizumab therapy, patients will have a brain MRI and if there is no evidence of disease progression, patients will receive 6 cycles of Bevacizumab and TMZ. Beginning a minimum of 28 days after the last radiation treatment the bevacizumab will be dosed at 10 mg/kg on day 1 and day 15 of each cycle. TMZ will be given at 150-200 mg/m2 qd on days 1-5 of each cycle. Each cycle is 28 days.
  Interventions: Drug: Bevacizumab; Drug: Temozolomide; Radiation: RT (Radiation Therapy)

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab will be administered at 10 mg/kg on day 1 and day 15. Four to six weeks following completion of concurrent IMRT, TMZ and bevacizumab, patients will receive 6 cycles of Bevacizumab.
  Other Names: Avastin
Drug: Temozolomide — Patients will be treated with hypofractionated IMRT (60 Gy in 10 Fx) and daily temozolomide at 75 mg/m2 qd concurrent with IMRT. Four to six weeks following completion of concurrent IMRT, TMZ and bevacizumab, temozolomide will be given at 150-200 mg/m2 qd on days 1-5 of each cycle.
  Other Names: Temodar
Radiation: RT (Radiation Therapy) — Patients will be treated with hypofractionated IMRT (60 Gy in 10 Fx)

SUMMARY:
The purpose of this study is to find out whether Hypofractionated Intensity-Modulated Radiation Therapy (Hypo-IMRT) combining with temozolomide chemotherapy can be safely given with a targeted agent, bevacizumab, and how effective this study treatment will be in controlling your brain tumor.

DETAILED DESCRIPTION:
This is a pilot phase II trial of the combination of concurrent hypofractionated IMRT (60 Gy/2 weeks), temozolomide and bevacizumab followed by 6 cycles of adjuvant bevacizumab and temozolomide in patients with grade IV malignant gliomas (glioblastoma and gliosarcoma). The study will have survival and toxicity endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of WHO grade IV primary malignant glioma (GBM or gliosarcoma).
* Age ≥ 18 years at the time of study registration
* Karnofsky Performance Scale ≥ 60%
* Absolute Neutrophil Count (ANC) ≥ 1,500 cells/mm3, hemoglobin ≥ 9.0 g/dl, platelets ≥ 100,000 cells/ mm3
* Serum creatinine ≤ 1.5 mg/dl, serum glutamate oxaloacetate transaminase (SGOT) and bilirubin ≤ 1.5 times upper limit of normal
* Signed informed consent approved by the Institutional Review Board
* Craniotomy or intracranial biopsy site must be adequately healed, free of drainage or cellulitis, and the underlying cranioplasty must appear intact at the time of study entry. Study treatment should be initiated > 28 days following the last surgical procedure (including open biopsy, surgical resection, wound revision, or any other major surgery involving entry into a body cavity)

Exclusion Criteria:

* Life expectancy of less than 12 weeks
* Prior treatment, including radiation therapy or chemotherapy, for GBM with the exception of surgery (Gliadel Wafers are allowed at the time of surgery)
* Active malignancy, with the exception of superficial basal cell and/or superficial squamous (skin) cell, or carcinoma in situ of the cervix
* Active infection requiring IV antibiotics
* Pregnant or breast feeding
* International normalized ratio (INR) > 1.5 and activated partial thromboplastin time (aPTT) > 1.5 × the upper limit of normal (ULN) (except for subjects receiving anticoagulation therapy) in the absence of therapeutic intent to anticoagulate the subject. Therapeutic anticoagulation is permitted
* Evidence of ≥ Common Toxicity Criteria for Adverse Effects (CTCAE) v.3 grade 2 CNS hemorrhage (CNS hemorrhage when medical intervention indicated), but grade 1 CNS hemorrhage (asymptomatic radiographic findings on the baseline brain CT or MRI only) is allowed. Punctate hemorrhage or the presence of hemosiderin is not considered a Grade 1 event for the purpose of this study. )
* Inadequately controlled hypertension (defined as systolic blood pressure >150 mmHg and/or diastolic blood pressure > 100 mmHg)
* Prior history of hypertensive crisis or hypertensive encephalopathy
* Current New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of myocardial infarction or unstable angina within 6 months prior to enrollment
* History of stroke or transient ischemic attack within 6 months prior to enrollment
* Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to enrollment
* History of hemoptysis (≥ 1/2 teaspoon of bright red blood per episode) within 1 month prior to enrollment
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to enrollment or anticipation of need for major surgical procedure during the course of the study
* Core needle biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to enrollment
* History of abdominal fistula or gastrointestinal perforation within 6 months prior to enrollment
* Serious, non-healing wound, active ulcer, or untreated bone fracture
* Proteinuria as demonstrated by a Urine protein-creatinine ratios (UPC) ratio ≥ 1.0 at screening (Appendix A).
* Known hypersensitivity to any component of bevacizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-09-16 (Actual); Primary Completion 2014-09-07 (Actual); Study Completion 2017-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Ney, M.D, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, University of Colorado Cancer Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RT With Temozolomide and Bevacizumab
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | RT With Temozolomide and Bevacizumab
Number analyzed (Participants) | 30
Age, Continuous [Mean (Full Range); unit: years] | 57 [31 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: 6-month Progression-free Survival
Description: To use 6-month progression-free survival to assess the efficacy of the combination of hypofractionated IMRT delivering 60 Gy over 2 weeks with concurrent bevacizumab and temozolomide followed by 6 cycles of adjuvant bevacizumab and temozolomide.
Time Frame: 6 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | RT With Temozolomide and Bevacizumab
Number analyzed (Participants) | 30
months | 90 [73.6 to 97.3]

2. Secondary Outcome: Overall Survival, Measured From the Day of Initial Diagnosis (Biopsy or Surgery) to the Time of Death From Any Cause.
Time Frame: follow up for life
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | RT With Temozolomide and Bevacizumab
Number analyzed (Participants) | 30
months | 16.3 [12.5 to 16.8]

ADVERSE EVENTS:
Arm/Group | RT With Temozolomide and Bevacizumab
Serious Adverse Events (participants affected / at risk) | 3/30
Other Adverse Events (participants affected / at risk) | 10/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RT With Temozolomide and Bevacizumab (N=30)
sepsis (Infections and infestations) | 1 (1)
cranial dehiscence/wound infection (Infections and infestations) | 1 (1)
seizure (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RT With Temozolomide and Bevacizumab (N=30)
myelosuppression (Blood and lymphatic system disorders) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No